CLINICAL TRIAL: NCT02499393
Title: Comparison of Two Method of Therapeutic Hypothermia Enhanced by Magnesium Sulphate in Neonatal Encephalopathy
Brief Title: Hypothermia Enhanced by Magnesium Sulphate
Acronym: Hemen
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Polish Mother Memorial Hospital Research Institute (Other)
Collaborators: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PolishMMHRI
Record Dates: First submitted 2015-07-01; First posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Perinatal Anoxic-ischemic Brain Injury
Keywords: newborn; therapeutic hypothermia; magnesium sulphate
MeSH Terms: interventions — Magnesium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TH+MgSO4 (Experimental): Therapeutic hypothermia plus magnesium sulphate intravenous infusion Neonates who were randomized to the study group (TH+MgSO4) received three 250 mg/kg doses of magnesium sulfate given as one - hour continuous infusion spaced 24 hours apart on three consecutive days. 20% Magnesium Sulfuricum (Polpharma), 2 g /10 ml were used.
  Interventions: Drug: Magnesium Sulfate
- TH- therapeutic hypothermia (No Intervention): therapeutic hypothermia without magnesium sulphate

INTERVENTIONS:
Drug: Magnesium Sulfate — intravenous infusion of magnesium sulphate
  Other Names: Magnesii Sulfurici 20% Polpharma
  Arms: TH+MgSO4

SUMMARY:
New 2010 neonatal resuscitation guidelines state that offering therapeutic hypothermia (TH) should be a standard of care in managing neonates with perinatal hypoxic - ischemic insult and present with signs of moderate and/or severe hypoxic - ischemic encephalopathy (HIE) . Despite the evidence from several randomized control trial (RCT) proving its effectiveness, its effect is perceived insufficient or only modest. Thus today's research efforts are directed toward finding the new possibilities of enhancing the effects of hypothermia. List of agents with potential neuroprotective properties includes: erythropoetin, melatonin, topiramate, morphine, xenon, MgSO4. Given investigators previous experiences with preterm neonates exposed to MgSO4 prenatally or administered this drug after birth because of perinatal asphyxia, the investigators designed the trial which would evaluate the possibility of increasing the TH effect by combining this method with MgSO4. Until now there are several published studies evaluating the effectiveness of MgSO4 in the group of asphyxiated neonates, including one RCT. However, all of these studies were conducted before the era of TH Furthermore, irrespective of the potential benefits, safety of using MgSO4 during TH in the group of term neonates was not studied. It is particularly important in the light of the results presented by Mittendorf et.al. They studied the effects of prenatal aggressive treatment with MgSO4 on the outcome of preterm neonates showed that patients exposed to high doses of MgSO4 were at higher risk of severe intracranial bleeding. Other side effects of high serum magnesium levels are: vasodilatation, hypotension, cardiac arrhythmias, coagulopathy, and gastrointestinal disturbances. MgSO4 is a very attractive neuroprotective option,also because of its easy availability. Drug can be administered in the birth hospital while neonate is being prepared for the transport to TH center. Timing of the intervention is very important for neonates suffering from perinatal asphyxia. Both TH and administration of potentially neuroprotective drug should be started during "therapeutic window". It is the initial potentially reversible phase of hypoxic insult lasting about 6 hours. If the long-term follow up shows that MgSO4 has an additive neuroprotective effect and no significant side effects in the group of asphyxiated neonates treated with TH this relatively simple and not expensive intervention may be introduced into clinical practice

DETAILED DESCRIPTION:
First decade of the twenty first century is an era when the therapeutic hypothermia became a widely used procedure in managing neonates with hypoxic - ischemic encephalopathy. New 2010 neonatal resuscitation guidelines state that offering therapeutic hypothermia should be a standard of care in managing neonates who sustained perinatal hypoxic - ischemic insult and present with signs of moderate and/or severe hypoxic - ischemic encephalopathy. Despite the evidence coming from several randomized controlled trials proving its effectiveness, in certain situations its effect is perceived insufficient or only modest at best. For this reason today's research efforts are directed toward finding the new possibilities of enhancing the effects of hypothermia. Some these new modalities are: modification of the hypothermia protocol, hypothermia combined with drugs which have a potential to be neuro-protective, and finally stem cell therapy. List of medications/substances with potential neuro - protective properties includes: erythropoetin, melatonin, topiramate, morphine, xenon, magnesium sulfate. Given investigators previous experiences with group of preterm neonates who were either exposed to magnesium sulfate prenatally or administered this drug after birth because of perinatal asphyxia, it was only natural to design the trial which would evaluate the possibility of increasing the effect of therapeutic hypothermia by combining this modality with administration of magnesium sulfate. Before the era of inhaled NO magnesium sulfate was widely used in the management of neonates with persistent pulmonary hypertension of neonates (PPHN), but then the level in the serum was kept in the high range (3,5 - 5,5 mmol/L). Until now there are several published studies evaluating the effectiveness of magnesium sulfate in the group of asphyxiated neonates, including one randomized controlled trial. Results are promising. However, all of these studies were conducted before the era of therapeutic hypothermia. Furthermore, irrespective of the potential benefits, safety of using magnesium sulfate during therapeutic hypothermia in the group of term and late preterm neonates was not studied. It is particularly important in the light of the results presented by Mittendorf et.al. They studied the effects of prenatal aggressive treatment with magnesium sulfate on the outcome of the neonates born with very low birth weight and showed that patients exposed to high doses of magnesium were at higher risk for developing severe intracranial bleeding. Other known side effects of high serum magnesium levels are: vasodilatation, hypotension, cardiac arrhythmias, coagulopathy, and gastrointestinal disturbances. Magnesium sulfate is a very attractive option as a neuroprotective drug also because of its easy availability. Drug can be administered to the patient in the birth hospital while neonate is being prepared for the transport to the center with therapeutic hypothermia. Timing of the intervention is very important in the management of the neonates suffering from perinatal asphyxia. Both, therapeutic hypothermia, as well as administration of potentially neuroprotective drug should be started during so called "therapeutic window". It is the initial potentially reversible phase of hypoxic insult lasting about 6 hours followed by the irreversible phase of apoptosis and destruction of neurons. If the long terms follow up shows that magnesium sulfate has an additive neuroprotective effect and no significant side effects in the group of asphyxiated neonates treated with therapeutic hypothermia this relatively simple and not expensive intervention may be introduced into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Group A Infants > 36.0 weeks gestation* with at least ONE of the following: * for gestational age also use clinical assessment

* Apgar score of less than or equal to ≤5 at 10 (ten) minutes after birth
* continued need for resuscitation, including endotracheal or mask ventilation, at 10min after birth
* acidosis defined as either umbilical cord pH or any arterial, venous or capillary pH within 60 min of birth less than (<) pH 7.00
* base deficit greater than or equal to (≥) 16 mmol/L in umbilical cord blood sample or any blood sample within 60 minutes of birth (arterial or venous blood)

Group B Newborn with moderate or severe encephalopathy with varying states of consciousness: lethargy, stupor, or coma and

One or more of below:

* hypotonia
* abnormal reflexes : oculomotor / pupillary
* suck: weak / absent
* clinical seizures - clinically confirmed

Group C integrated electroencephalogram (aEEG / CFM) (lasting at least 20 minutes), which indicates either a moderate / serious abnormalities in the background activity aEEG (a score of 2 or 3) or convulsions attacks.

Exclusion Criteria:

* major congenital maformation
* extremely poor prognosis : Apgar score 0 @ 15 minutes of life

Ages: 1 Hour to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2010-04; Primary Completion 2013-04 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Death | until discharge (participants will be followed for the duration of hospital stay @ hypothermia center, an expected up to 4 weeks

SECONDARY OUTCOMES:
Neurological status | 1-7 DOL
  according to Thompson scale (Hypoxic-ischemic encephalopathy score)
Neurological status | 24 months
  the long-term evaluation of psychomotor development according to the scale BAYLEY III

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Gulczynska, MD PhD, Principal Investigator — Polish Mother Memorial Hospital Research Instutute
Locations (1):
- Polish Mother Memorial Hospital - Research Instutiute, Lodz, Poland

REFERENCES:
- [Background] Merchant N, Azzopardi D. Early predictors of outcome in infants treated with hypothermia for hypoxic-ischaemic encephalopathy. Dev Med Child Neurol. 2015 Apr;57 Suppl 3:8-16. doi: 10.1111/dmcn.12726. PMID 25800487
- [Derived] Gulczynska EM, Gadzinowski J, Kesiak M, Sobolewska B, Caputa J, Maczko A, Walas W, Cedrowska-Adamus W, Talar T. Therapeutic hypothermia in asphyxiated newborns: selective head cooling vs. whole body cooling - comparison of short term outcomes. Ginekol Pol. 2019;90(7):403-410. doi: 10.5603/GP.2019.0069. PMID 31392710